CLINICAL TRIAL: NCT01082263
Title: Midazolam Drug-Drug Interaction Study With Lurasidone HCl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1050269
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Schizophrenia Patients
Keywords: DDI study between Midazolam and Lurasidone HCl; Male and Female
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midazolam/Lurasidone (Other): Schizophrenia patient
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — Day1: 5 mg midazolam (2.5 mL of the 2 mg/mL syrup) Day6: 120 mg lurasidone (three 40 mg tablets) + 5 mg midazolam (2.5 mL of the 2 mg/mL syrup) Day 7-12: 120 mg lurasidone (three 40 mg tablets) 120 mg lurasidone (three 40 mg tablets) on Day 13 + 5 mg midazolam (2.5 mL of the 2 mg/mL syrup)

SUMMARY:
A Phase I, Drug-Drug Interaction Study between Midazolam and Lurasidone HCl.

DETAILED DESCRIPTION:
lurasidone 120 mg, midazolam 5 mg

To compare the single-dose pharmacokinetic profile of midazolam 5 mg when administered alone vs. when administered with a single-dose of lurasidone 120 mg.

To compare the single dose pharmacokinetic profile of midazolam 5 mg when administered alone vs. when administered after steady state dosing with lurasidone 120 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorders
2. Females who participate in this study:

   are unable to have children -OR- are willing to remain abstinent from Day -5 to 90 days after discharge; -OR- are willing to use an effective method of double-barrier birth control from Day -5 to 90 days after discharge.
3. Males must be willing to remain sexually abstinent or use an effective method of birth control from Day -5 to 90 days after discharge.
4. Able and agree to remain off of prior antipsychotic medication for the duration of the study.

Exclusion Criteria:

1. Known presence or history of renal or hepatic insufficiency.
2. A history or presence of abnormal electrocardiogram (ECG5. Known history or presence of clinically significant intolerance to antipsychotic medications.
3. Significant orthostatic hypotension (i.e. a drop in systolic blood pressure of 30 mmHg or more and/or drop in diastolic blood pressure of 20 mmHg or more on standing).
4. Presence or history (within the last year) of a medical or surgical condition (e.g. gastrointestinal disease) that might interfere with the absorption, metabolism, or excretion of orally administered lurasidone.
5. Participated in another clinical trial or receiving an investigational product within 30 days prior to drug administration.
6. Use of concomitant medications that prolong the QT/QTc interval within 14 days prior to Day -5 to follow-up including but not limited to those listed in Appendix 19.5.
7. Received depot neuroleptics unless the last injection was at least 1 treatment cycle before Day -5.
8. Difficulty fasting or consuming the FDA high fat meals.
9. At risk with midazolam dosing with respiratory disease or impaired gag reflex, in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Bussel, MD, Principal Investigator — CCT/Parexel
Locations (1):
- CCT/Parexel, Culver City, California, United States